CLINICAL TRIAL: NCT03093077
Title: Kinematics Following Total Knee Arthroplasty Performed With Different Surgical Alignment Techniques
Brief Title: Kinematics After Total Knee Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unanswered questions regarding indications for device.
Sponsor: Kristin Zhao, PhD (Other)
Responsible Party: Sponsor-Investigator, Kristin Zhao, PhD, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15-008300
Record Dates: First submitted 2016-09-26; First posted 2017-03-28 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anatomic alignment (Experimental): The aim of anatomic alignment is to recreate an individual's pre-operative alignment using the DePuy ATTUNE total knee arthroplasty system.
  Interventions: Device: DePuy ATTUNE total knee arthroplasty system
- Mechanical alignment (Active Comparator): The aim of mechanical alignment is to achieve a neutral mechanical alignment regardless of pre-operative status, using the DePuy ATTUNE total knee arthroplasty system.
  Interventions: Device: DePuy ATTUNE total knee arthroplasty system

INTERVENTIONS:
Device: DePuy ATTUNE total knee arthroplasty system — A standard midvastus approach will be used for both alignment technique groups. This is a standard approach for exposing the knee joint for TKA.

SUMMARY:
The purpose of this study is to evaluate and compare implant kinematics of conventional mechanically aligned and anatomically aligned total knee arthroplasties (TKA) at 1 year post-operatively.

DETAILED DESCRIPTION:
Participants will be randomized to receive a primary TKA using either an anatomic alignment or a conventional mechanical alignment technique.

Participants will undergo a kinematic analysis of a deep knee bend using single-plane fluoroscopy at 1 year post-operatively. The primary outcome will be based on the 6 degree of freedom kinematics and associated joint component proximity during the knee bend task. Secondary outcomes include the Knee Society Score, the Knee Injury and Osteoarthritis Outcome Score, and the Forgotten Knee Score.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Primary arthroplasty for treatment of osteoarthritis
* Age between 40 and 80 years old
* Willingness to provide written consent for study participation

Exclusion Criteria:

* Revision arthroplasty
* Pre-operative knee flexion lower than 90 degrees
* Varus knee deformity greater than 15 degrees
* Pre-operative valgus knee deformity
* Presence of infections, highly communicable diseases or metastatic disease
* Significant neurological or musculoskeletal disorders or disease that may interfere with normal gait or weight bearing
* Congenital, developmental, or other bone disease or previous hip surgery that may, in the surgeon's judgment, interfere with total knee prosthesis survival or success
* Presence of previous prosthetic knee or hip replacement device
* BMI > 40
* Pregnant women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Knee motion, as determined by 6 degree freedom of movement kinematics and associated joint proximity during the knee bend task. | 1 year post surgery

SECONDARY OUTCOMES:
Participants perception of knee function, as determined by the Knee injury Osteoarthritis Outcome Score (KOOS) | 1 year post surgery
Participant's awareness of the joint implant, as determined by the Forgotten Joint Score (FJS-12) | 1 year post surgery
Knee joint and ambulatory function based on physical exam, as determined by the Knee Society Score (KSS) | 1 year post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kristin D. Zhao, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided